CLINICAL TRIAL: NCT01522807
Title: A Phase I, Cross-Over, Single Dose, Double-Blind Study To Estimate The Relative Bioavailability Of Three Different Formulations Of PF-05190457 In Healthy Adult Volunteers
Brief Title: A Study Of Three PF-05190457 Formulations In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: B3301007
Record Dates: First submitted 2011-10-30; First posted 2012-02-01 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Phase 1; Single Doses; Biocomparison; Pharmacokinetics; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — PF-5190457

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 100 mg PF-05190457 (Experimental): Three fasted treatments and fed with the short-duration osmotic capsule
  Interventions: Drug: PF-05190457
- 100 mg PF - 05190457 (Experimental): Three fasted treatments and fed with the long-duration osmotic capsule
  Interventions: Drug: PF-05190457

INTERVENTIONS:
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a suspension in the fasted state
  Arms: 100 mg PF-05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a short-duration osmotic capsule in the fasted state
  Arms: 100 mg PF-05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a long-duration osmotic capsule in the fasted state
  Arms: 100 mg PF-05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a short-duration osmotic capsule in the fed state
  Arms: 100 mg PF-05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a suspension in the fasted state
  Arms: 100 mg PF - 05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a short-duration osmotic capsule in the fasted state
  Arms: 100 mg PF - 05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a long-duration osmotic capsule in the fasted state
  Arms: 100 mg PF - 05190457
Drug: PF-05190457 — 100 mg single oral dose of PF-05190457 is administered as a long-duration osmotic capsule in the fed state
  Arms: 100 mg PF - 05190457

SUMMARY:
The purpose of the study is to evaluate the plasma drug concentrations of three formulations of PF-05190457 after administration of single doses to healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females of non-childbearing potential between ages of 21 and 55 years, BMI of 17.5 to 30.5 kg/m^2, and weight above 50 kg.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2011-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
The single dose pharmacokinetics of PF-05190457 in three formulations will be described by estimating parameters of Area Under the Curve (AUC) and its ratio between formulations as data permit. | 0 - 48 hours post dose
The single dose pharmacokinetics of PF-05190457 in three formulations will be described by estimating parameters of Maximum Concentration (Cmax) and its ratio between formulations as data permit. | 0 - 48 hours post dose
The single dose pharmacokinetics of PF-05190457 in three formulations will be described by estimating parameter of Time of Maximum concentration (Tmax) as data permit. | 0 - 48 hours post dose
The single dose pharmacokinetics of PF-05190457 in three formulations will be described by estimating parameter of Elimination of half-life (t ½ ) as data permit. | 0 - 48 hours post dose

SECONDARY OUTCOMES:
The ratio of fasted to fed single dose pharmacokinetics of PF-05190457 in two test formulations will be described by estimating parameters of Area Under the Curve (AUC) and its ratio between fed states as data permit. | 0 - 48 hours post dose
The ratio of fasted to fed single dose pharmacokinetics of PF-05190457 in two test formulations will be described by estimating parameters of Maximum Concentration (Cmax) and its ratio between fed states as data permit. | 0 - 48 hours post dose
Changes in plasma glucose and insulin due to single doses of three formulations of PF-05190457 will be estimated. | 0 - 24 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3301007&StudyName=A%20Study%20Of%20Three%20PF-05190457%20Formulations%20In%20Healthy%20Volunteers